CLINICAL TRIAL: NCT04649697
Title: Evaluation of Topical Rebamipide Versus Topical Clobetasol in Management of Methotrexate-Induced Oral Ulceration in Rheumatoid Arthritis Patients: Randomized-Controlled Clinical Trial
Brief Title: Rebamipide (Regular & Nanoparticulated) vs. Clobetasol in Management of Methotrexate-Induced Oral Ulceration in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Abd el-Aziz Mohamed, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBC-CU-2020-9
Record Dates: First submitted 2020-10-26; First posted 2020-12-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rebamipide; Clobetasol; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rebamipide (Experimental): The enrolled subjects will be treated with Rebamipide in mucoadhesive gel for 2 weeks or until complete healing.
  Interventions: Drug: Rebamipide
- Nanoparticulated Rebamipide (Experimental): The enrolled subjects will be treated with nanoparticulated Rebamipide in mucoadhesive gel for 2 weeks or until complete healing.
  Interventions: Drug: Nanoparticulated Rebamipide
- Clobetasol (Active Comparator): The enrolled subjects will be treated with Clobetasol in mucoadhesive gel for 2 weeks or until complete healing.
  Interventions: Drug: Clobetasol Propionate

INTERVENTIONS:
Drug: Rebamipide — A mucosal protection drug developed in Japan for the treatment of gastritis and gastric ulcer.
  Other Names: Mucosta
  Arms: Rebamipide
Drug: Nanoparticulated Rebamipide — A mucosal protection drug developed in Japan for the treatment of gastritis and gastric ulcer will be used in nanotechnology.
  Other Names: Mucosta
  Arms: Nanoparticulated Rebamipide
Drug: Clobetasol Propionate — A corticosteroid drug used as a gold standard for treatment of methotrexate induced oral ulceration.
  Other Names: corticosteroids
  Arms: Clobetasol

SUMMARY:
The aim of this intervention study is to compare the effect of topical Rebamipide (regular and nanoparticulated) to topical Clobetasol propionate in management of Methotrexate induced oral mucositis in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
A random sample of patients diagnosed with rheumatoid arthritis attending at the Rheumatology clinic in faculty of Medicine, Cairo University Hospital, will be enrolled by the investigator in the study in a consecutive order after being examined for methotrexate induced oral ulceration by means of history and clinical examination.

Since oral mucositis associated with Methotrexate include production of free radicals, increase of inflammatory cytokines, and alteration of intracellular signal transduction, this suggests that Rebamipide should be useful for its treatment and prevention. Thus, this RCT will be the first to evaluate the treatment of Methotrexate-induced oral mucositis using Rebamipide and Rebamipide nanoparticles in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient who agreed to sign the informed consent.
* Age: 20-70 years old.
* Gender: males and females
* RA patients treated with MTX and suffering from MTX-induced oral ulceration.

Exclusion Criteria:

* Patients refused to sign the informed consent.
* Pregnant or lactating females in their child bearing age group.
* patients with known or suspected history of hypersensitivity to any of the ingredients of the preparation of the drugs used.
* Systemic disease: such as uncontrolled diabetes mellitus, auto-immune diseases known to cause oral ulceration, renal or liver dysfunction or any other condition considered risky by the clinician.
* Patients treated with any medication for the condition at the time of setting.
* Salivary gland diseases.
* Malignancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
change in the Clinical improvement of oral ulcers | assessment will be at baseline, 2 weeks and 4 weeks
  Will be assessed using World Health Organization (WHO) grading of mucositis

SECONDARY OUTCOMES:
Subjective degree of pain | Pain assessment will be daily for the first week then at 2 weeks and 4 weeks.
  All patients were introduced to the Numerical Rating Scale (NRS) and learnt how to express their pain through it, patients were instructed to fill the scale paper at the first visit [baseline], this procedure was repeated for each follow-up visit.
size of oral ulcer | assessment at 0, 2 weeks and 4 weeks
  The ulcer size was determined by measuring the distance between two opposite edges of the ulcer border, using a periodontal probe in millimeters.
healing time of the ulcer | assessment at 0, 2 weeks and 4 weeks
  The total healing time of oral ulcers Will be recorded in days for all the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt